CLINICAL TRIAL: NCT06128642
Title: Comparison of the Effects of Two Different Orthoses on Individuals With Hallux Valgus
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, sena ozdemir, Assistant Prof., Istanbul Medipol University Hospital
Other Study IDs: MedipolUniversity
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Hallux Valgus
Keywords: Dynamic orthosis; Toe separator orthosis; Hallux valgus angle; Plantar pressure analysis; orthosis satisfaction
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Toe separator orthosis: The silicone toe spreader orthosis does not use tape or straps to separate the first and second toes and pull them medially to realign the first metatarsal. Orthotics reduce the pain in the bunion area by reducing the high friction between the shoe and the bunion. Participants will be asked to use their orthoses for an average of 8 hours per day for 1 month.
  Interventions: Device: Toe separator orthosis
- Dynamİc orthosis: The dynamic orthosis contains a free joint that does not hinder the movement of the first metatarsophalangeal joint. The working principle of the orthosis is to provide healing of the deformity with low torque and long-term stretching. The dynamic orthosis corrects the hallux valgus angle by realigning the hallux, thus allowing plantarflexion and dorsiflexion. Participants will be asked to use their orthoses for an average of 8 hours per day for 1 month.
  Interventions: Device: Dynamic orthosis

INTERVENTIONS:
Device: Toe separator orthosis — The orthoses to be used during the study will be randomly distributed to the individuals participating in the study. Foot pressure analysis will be evaluated after the participants use the toe separation orthosis for 8 hours a day, for a total of 1 month.
  Plantar pressure analysis will be performed again without orthosis, with orthosis and 1 month after the use of orthosis. Additionally, patient orthosis satisfaction evaluation will be made at the end of the 1-month period during which the participants use the orthoses.
  Groups: Toe separator orthosis
Device: Dynamic orthosis — The orthoses to be used during the study will be randomly distributed to the individuals participating in the study. Foot pressure analysis will be evaluated after participants use the dynamic orthosis for 8 hours a day, for a total of 1 month.
  Plantar pressure analysis will be performed again without orthosis, with orthosis and 1 month after the use of orthosis. Additionally, patient orthosis satisfaction evaluation will be made at the end of the 1-month period during which the participants use the orthoses.
  Groups: Dynamİc orthosis

SUMMARY:
Hallux valgus (HV) is a tri-planar, painful and common foot deformity characterized by the medial orientation of the first metatarsal, lateral deviation and pronation of the big toe at the level of the first metatarsophalangeal joint. Due to the increase in the severity of hallux valgus deformity, dissatisfaction with the appearance of the foot, difficulty choosing shoes due to bunions and pain, difficulty walking and accordingly, restriction in daily activities, the functional levels and health-related quality of life of individuals are negatively affected. The aim of this study is to compare the effect of using a toe separator orthosis and dynamic orthosis for 1 month on hallux valgus angle and plantar pressure in individuals with hallux valgus.

DETAILED DESCRIPTION:
If left untreated, hallux valgus becomes a painful and progressive disease of the big toe that severely restricts the patient's daily activities and disrupts the aesthetic appearance of the foot. As the deformity progresses, dissatisfaction with the appearance of the foot, difficulty in choosing shoes, difficulty in walking and, accordingly, limitation in daily activities, arch pathologies Individuals' health-related quality of life and functional levels are negatively affected due to problems such as nail problems, bunions and callus formations.

Surgical and conservative treatment methods are used in the treatment of hallux valgus deformity. Conservative treatment methods are more preferred due to possible complications of surgical treatment methods such as infection, skin problems, bone nonunion, bone malunion, hallux valgus and complex regional pain syndrome. Conservative treatment methods aim to reduce the hallux valgus angle (HVA) in individuals with hallux valgus deformity, reduce pain and prevent the severity of the deformity from increasing.

Different orthosis applications are used in the conservative treatment of hallux valgus deformity. In the literature, it is reported that finger spreader orthosis, dynamic orthosis, and night orthosis are effective in the treatment of mild and moderate hallux valgus deformities. The most commonly used finger separator orthoses and dynamic orthoses in clinics are orthoses with proven effectiveness in the treatment of hallux valgus deformity, but there is no study comparing the effectiveness of these orthoses. The purpose of this study is to examine the effect of toe separation orthosis and dynamic orthosis on hallux valgus angle and plantar pressure.

The individuals included in the study will be randomly divided into two groups: those using the finger separation orthosis and those using the dynamic orthosis.

Foot pressure analysis after the participants use the toe separation orthosis and dynamic orthosis for 1 month will be evaluated. Pressure analysis evaluation will be performed 3 times; before using the orthosis, when first wearing the orthosis, and 1 month after using the orthosis.

Individuals participating in the study must first sign the informed consent form. Individuals who agree to participate in the study will fill out the socio-demographic evaluation form.

According to the Manchester Scale, the individual's hallux valgus deformity will be classified according to its severity.

Hallux valgus angle measurement will be made with a goniometer. In order to understand the effect of deformity on individuals, the Foot Function Index Evaluation Form will be filled out by individuals. For the pain, function and alignment evaluation of individuals, the evaluation form prepared by the American Orthopedic Foot-Ankle Society (AOFAS) will be answered by individuals. The Manchester-Oxford foot questionnaire will be administered to assess standing, walking and quality of life.

The orthoses to be used during the study will be randomly distributed to the individuals participating in the study. Plantar pressure analysis will be performed without orthosis, with orthosis and 1 month after the use of orthosis. At the end of the 1-month period during which individuals use the orthoses, patient orthosis satisfaction will be evaluated.

Socio-Demographic evaluation will include physical evaluations such as individuals' name, surname, age, weight and body mass index. For social evaluation, individuals' education level, profession and job status will be asked. Questions that are important for the research are included in the socio-demographic evaluation. For this study, individuals will be asked about their shoe choice, average number of steps per day, average standing time per day, presence of hallux valgus, and presence of hallux valgus in the family. Additionally, the foot will be evaluated and the presence of pes planus will be examined.

It is a scale developed by Garrow to classify hallux valgus deformity. It deals with hallux valgus deformity at 4 levels; none (1), mild (2), moderate (3), severe (4). The classification is evaluated by comparing 4 different photographs containing the hallux valgus deformity between individuals with the deformity.

A universal standard goniometer will be used to measure the hallux valgus angle. To measure the hallux valgus angle, the pivot part of the goniometer is placed in the 1st Metatarsophalangeal joint. One arm of the goniometer is placed parallel to the 1st Metatarsal bone and the other arm is parallel to the proximal phalanx, the angle between them is measured and the hallux valgus angle is found. Hallux valgus angle is classified as normal (<15°), mild (15-20°), moderate (20°-40°) and severe (>40°).

Foot function index is a widely used form that can be filled out by the person himself, developed to measure the effects of foot pathologies on pain, disability and activity limitation.

Foot function index is used in research on children, adults and older adults to determine the effectiveness of treatment for various foot and ankle problems such as congenital, acute and chronic diseases and injuries, as well as after surgical interventions or orthosis use.

Foot function index; It consists of 23 items with 3 subgroups: pain, disability and activity limitation. While the nine-item pain subscale measures the level of foot pain in various situations, the 9-item disability subscale determines the degree of difficulty in performing various functional activities due to foot problems. With the activity limitation subscale, which includes five items, activity limitations due to foot problems are evaluated.Foot function index is a widely used form that can be filled out by the person himself, developed to measure the effects of foot pathologies on pain, disability and activity limitation.

Foot function index is used in research on children, adults and older adults to determine the effectiveness of treatment for various foot and ankle problems such as congenital, acute and chronic diseases and injuries, as well as after surgical interventions or orthosis use.

Foot function index; It consists of 23 items with 3 subgroups: pain, disability and activity limitation. While the nine-item pain subscale measures the level of foot pain in various situations, the 9-item disability subscale determines the degree of difficulty in performing various functional activities due to foot problems. With the activity limitation subscale, which includes five items, activity limitations due to foot problems are evaluated. Patients score all items with the Visual Analogue Scale (VAS), taking into account their foot conditions one week ago. To calculate the subscales and total score, the scores of each item are summed, divided by the sum of the maximum scores of the items and multiplied by 100. Higher scores indicate greater pain, disability, and activity limitation. Turkish validity study was conducted.

American Orthopedics Foot and Ankle Society (AOFAS); Separate scales were created for four different parts of the foot; The ankle-hindfoot scale (AHFS) is a scale for the midfoot, a scale for the metatarsophalangeal and interphalangeal joints of the hallux (AOFAS-MTF-IF), and a scale for the metatarsophalangeal and interphalangeal joints of the other toes, allowing their application to different types of injuries and treatments. For this study, function, pain and alignment will also be evaluated with the AOFAS-MTF-IF scale. Pain is evaluated over 40 points, function is evaluated over 45 points, and alignment is evaluated over 15 points. A total of 100 points are collected in the evaluation. While low scores indicate poor prognosis, high scores indicate good prognosis. Turkish validity study was conducted.

The Manchester-Oxford Foot Questionnaire (MOXFQ) is a practical, valid and reliable questionnaire that accurately assesses patients with hallux valgus. The MOXFQ is a recently designed, patient-reported outcome measure developed with patients so that it adequately records their perception of their symptoms. Accordingly, MOXFQ is a suitable scale for evaluating the functional and social effects of individuals with hallux valgus on walking, standing and quality of life, as well as pain. This questionnaire is therefore very useful and can be used in clinical trials and for comparison between groups undergoing different treatment options. Turkish validity study was conducted.

To measure the pressure distribution during walking, it will be done with the Sensor Medica brand, which is the plantar pressure measurement system within the Prosthesis / Orthosis Center (POMER) at Istanbul Medipol University. Free Step software compatible with the device will be used during pressure measurement.

Plantar pressure analysis refers to the measurement of the magnitude and distribution of the force applied to the plantar surface of the foot during walking. Plantar pressure analysis will be performed with the Sensor Medica device, which consists of pressure-sensitive sensors. Participants will wear socks during pressure measurement. Plantar pressure analysis will be performed on the participants 3 (three) times: without orthosis, when wearing the orthosis for the first time and 1 (one) month after using the orthosis.

To measure orthosis satisfaction after orthosis use, orthosis quality, comfort in orthosis use, difficulty of putting on and taking off, and suitability of the material will be evaluated. After using the orthosis, participants will evaluate these parameters with scores from 0 to 10. A score of 0 indicates that they are not at all satisfied with the orthosis, 5 points indicate neutral status, and 10 points indicate that they are very satisfied with the orthosis. Participants will express orthosis satisfaction by scoring the parameters in this way.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* Having mild to moderate hallux valgus deformity.

Exclusion Criteria:

* Individuals have cognitive, mental or psychological problems,
* Having previously used orthosis treatment for hallux valgus,
* Having a history of surgery on the foot,
* Presence of rheumatoid arthritis disease,
* Hallux valgus deformity is rigid.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To determine the participants, it is planned to prepare a poster with the visual of hallux valgus deformity, create it in physical forms, hang it on notice boards and share it online. Volunteers who want to participate in the study will be contacted and invited to be evaluated. Participants who meet the inclusion and exclusion criteria determined in the study will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Hallux valgus angle | 2 minute
  A goniometer will be used to measure the participants' degree of hallux valgus. Hallux valgus measurement of all participants will be performed by a single researcher.
  In measurement with goniometer; The hallux valgus angle will be obtained by placing the pivot part of the goniometer on the participant's foot parallel to the metatarsophalangeal joint, one arm parallel to the first metatarsophalangeal joint and the other parallel to the proximal phalanx, and measuring the angle between them.
Plantar pressure | 2 minute
  To measure the pressure distribution of the participants, the Sensor Medica device, the Free Step software compatible with the device will be used.
  The platform of the device is the FreeMed Maxi Baropodometric Platform. It is a pedobarographic evaluation device with a size of 60x50 cm, made of platform aluminum, capable of measuring a maximum pressure of 150 N/cm², with 2.5 dpi XY, 8 bit Z resolution, 3,000 sensors, and a sensor life of 1,000,000 cycles. In our study, static pressure analysis will be performed. During the analysis, the individual will be asked to stand on the platform facing forward, press the 'start' button in the program while his eyes are open on the platform as specified, and the patient will be asked to stand on the platform for 5 seconds without moving.
  Within the scope of static analysis measurements; Left-right forefoot, hindfoot and total foot loading percentages, left-right forefoot, hindfoot weight ratio percentage data will be recorded.

SECONDARY OUTCOMES:
Foot Questionnaire | 5 minute
  The Manchester-Oxford Foot Questionnaire (MOXFQ) is a recently designed, patient-reported outcome measure developed with patients so that it adequately records their perception of their symptoms. Accordingly, MOXFQ is a suitable scale for evaluating the functional and social effects of individuals with hallux valgus on walking, standing and quality of life, as well as pain.
  MOXFQ consists of 3 subheadings that are scored separately; It consists of a total of 16 questions: foot pain (5 questions), walking and standing (7 questions), and social interaction (4 questions). Each of the questions has 5 different answer options and is scored between 0-4, with 4 points representing a very severe situation. The score for each subheading ranges from 0 to 100; A score of 0 indicates the best possible clinical situation, and a score of 100 indicates the worst possible situation.
Evaluation of orthosis satisfaction | It takes the participant a maximum of 2 minutes to fill out the form.
  A satisfaction evaluation will be made for the participants in the study after using the hallux valgus orthosis. The numerical evaluation created by us will be used to evaluate the participants' orthosis satisfaction. The parameters evaluated in orthosis satisfaction are orthosis quality, comfort in using the orthosis, difficulty of wearing and removing it, and suitability of the material. After using the orthosis, participants will evaluate these parameters with scores from 0 to 5. A score of 0 indicates that you are not at all satisfied with the orthosis, 3 points indicate neutral status, and 5 points indicate that you are very satisfied with the orthosis. Participants will evaluate orthosis satisfaction by scoring the parameters in this way.

CONTACTS AND LOCATIONS:
Overall Officials: SENA ÖZDEMİR GÖRGÜ, PhD, Principal Investigator — Istanbul Medipol Universty
Locations (1):
- Sena Özdemir Görgü, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Camur H, Ozdemir Gorgu S. Comparison of the effects of orthoses on hallux valgus angle and plantar pressure in individuals with hallux valgus. Prosthet Orthot Int. 2025 Oct 1;49(5):494-501. doi: 10.1097/PXR.0000000000000423. Epub 2024 Dec 24. PMID 39721066